CLINICAL TRIAL: NCT02451644
Title: The Association Between Physical Activity and Pregnancy Rate Following Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Shalom Mazaki-Tovi MD, Director of high risk Department, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2043-15-SMC
Record Dates: First submitted 2015-05-09; First posted 2015-05-22 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- high risk for PTD with pedometer (Experimental): Patient with high risk for preterm delivery including short cervix or rapture of membranes
  Interventions: Device: pedometer

INTERVENTIONS:
Device: pedometer — patient will cary pedometer

SUMMARY:
The study examines the association between the amount of physical activity of the patient, ie the number of steps daily / weekly, and the pregnancy rate after embryo transfer.

DETAILED DESCRIPTION:
Many studies have investigated the matter until today and still no reliable information about the relationship between physical activity and / or its intensity and the pregnancy rate after embryo transfer.

All patients that would take part in the study will be given a pedometer to measure steps for a month.

Measuring steps will begin preparation for embryo transfer and two weeks after. Collected information about pregnancy rate (BHCG positive or negative).

ELIGIBILITY:
Inclusion Criteria:

* Participant speaks Hebrew or English speakers
* The participant is eligible to legally provide informed consent

Exclusion Criteria:

* The Subject in the wheelchair-bound or limited walking
* Participant refuses to give informed consent

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Physical activity as assessed by number of steps recorded by pedometer | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shalom Mazaki tovi, Ramat Gan, Israel